CLINICAL TRIAL: NCT06855901
Title: Home Ultra-longterm EEG Monitoring for Rare Epilepsies and Developmental and Epileptic Encephalopathies. an Open Label Nonpharmacological Interventional Prospective Study by Means of Minimally Invasive Wearable EEG Device
Brief Title: Home Ultra-long Term EEG Monitoring for Rare Epilepsies and Developmental and Epileptic Encephalopathies
Acronym: EMIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Collaborators: Azienda Ospedaliera Universitaria Federico II (AOU Federico II) (Unknown); Azienda Sanitaria Universitaria Giuliano Isontina [ASUGI], Università di Trieste, Italy (Unknown); Ospedale Pediatrico Bambino Gesù, Rome (IT) (Unknown)
Responsible Party: Principal Investigator, Stefano Meletti, MD, PhD, Azienda Ospedaliero-Universitaria di Modena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PNRR-MR1-2022-12376491; 33/2023/DISP/AOUMO (Other: AOU MO - Ministero della Salute); 127/2023/DISP/AOUMO (Other: AOU MO - Ministero della Salute)
Record Dates: First submitted 2025-02-22; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Epilepsies; Epilepsies, Focal; Epileptic Encephalopathy
Keywords: Epilepsy; Epileptic encephalopathies; subscalp EEG; Ultra-long EEG monitoring
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Group (Experimental): Patients with drug-resistant epilepsies. Age > 12 years
  Interventions: Device: Ultra-longterm EEG monitoring at home by means of a scubscalp electrode implant.

INTERVENTIONS:
Device: Ultra-longterm EEG monitoring at home by means of a scubscalp electrode implant. — Subjects with uncontrolled seizures previously investigated in outpatients epilepsy clinics and for whom an admission to the Epilepsy Monitoring Unit is indicated by clinical practice, will be screened for eligibility.
  Implantation of subcutaneous EEG electrodes will be done at each Research Unit by a neurosurgeon/surgeon. The implantation procedure will consist of placing subcutaneously the electrode contacts over the site of the suspected seizure focus as defined by a previous Video-EEG and neuroimaging evaluations. Surgical procedures will be performed under local anesthesia. If the device is well-tolerated, all the subjects will proceed to the extended home monitoring study, which is the core of the study protocol. The aim of the extended study is to assess sensitivity of seizure detection of sqEEG in comparison to subject's home diary, and the tolerability and safety of sqEEG in a period of 6 months.
  Other Names: EEG SubQ subcutaneous EEG device

SUMMARY:
With this study the Investigator expects to develop a precise patient-centered model of care by means of home ultra-long-term EEG monitoring with a minimally invasive wearable EEG device (sqEEG).

The following aims will be pursued:

1. to assess the sensitivity, reliability, and safety of sqEEG to record seizures over prolonged periods;
2. to verify sensitivity and reliability of automated seizure detection algorithms and to assess circadian and ultradian seizure/interictal epileptic discharges; distribution for the development of personalized seizure action plan;
3. to evaluate whether data collected with sqEEG can improve the clinical management of the patients and treatment outcomes.

The investigator expects to use this wearable at-home EEG device to obtain an objective quantification of electrographic and electro-clinical seizures over a twelve-week period up to twenty-four weeks at home. The precise quantification of seizures is essential for a tailored treatment approach and to effectively monitor the response to treatment adjustments.

The potential innovation of this approach relies on the possibility of managing the patient at home, reducing the side effects related to hospitalization and objectively quantifying the disease burden in the real-life setting with the aim of improve globally the patients' quality of life.

DETAILED DESCRIPTION:
Initial screening of the subjects.

Subjects with DEE or rare epilepsies with uncontrolled seizures and previously investigated in outpatients epilepsy clinics and in the Epilepsy Monitoring Unit (EMU) will be evaluated by review of the medical records.

The aim is to select subjects in whom assessment of seizure frequency is extremely relevant for their clinical management, including adjustment of medicines and need of support measures in their daily life. The indication to recruit also patients with epilepsy and intellectual disabilities is supported by the evidence that in these patients, either when living at home or in institutions, it is particularly difficult to have an objective assessment of their seizure frequency and of the response to treatment or to treatment adjustments. The use of sqEEG in this group of patients is therefore expected to provide extremely valuable information on the disease severity (i.e. seizure frequency) and the epilepsy modification following treatment changes.

The subjects will be selected regardless of a diagnosis of focal or generalized epilepsy, and regardless previous surgical treatments.

Recruitment and consent. The written consent form will be presented and discussed with the subject/legal guardians; all questions related to the informed consent will be answered. In all cases patients will receive detailed information regarding the procedure and purposes.

Study plan The project design includes two sequential parts, 'Part 1' which is a short-term study evaluating sqEEG compared to standard EEG monitoring. 'Part 2' represent the core of the project and consists of the ultra-longterm sqEEG monitoring at home for at least 12 weeks (up to 24 weeks).

Study Part 1:

* Subjects selection and recruitment
* Implantation of subcutaneous EEG electrodes by a surgeon/neurosurgeon. The implantation procedure will take care to place subcutaneously the electrode contacts over the site of the seizure focus as defined by a previous epilepsy data of the patients. The implantation will be unilateral in case of documented unilateral ictal epileptic discharges, or generalized epilepsies. In patients with independent bilateral seizure onset the implant will be bilateral.
* Earliest 10 days after the surgical procedure, the subjects will be admitted to the EMU as part of clinical practice activity at the investigational site, with the aim of recording their seizures both with video-EEG and sqEEG. This will allow the Neurologist:

  1. to test the sensitivity of sqEEG to detect seizures as compared to video-EEG (standard procedure);
  2. to assess the rate of false positives (FP) and false negatives (FN) detections
  3. to test the tolerability of sqEEG in the short term;
  4. to test the algorithm for automatic seizure detection in this initial set of EEG data;
  5. to test the safety of the sqEEG in the short term;
* Admission in EMU will last from 2 days to 2 weeks based on the number of seizures recorded (one electrographic or electroclinical seizure recorded on scalp EEG is advisable). At the end of EMU admission, seizure identification and quantification will be performed independently by the personnel of EMU and by the reviewer of sqEEG data. Both will be blinded of each other's results. Then the results will be compared.

Study Part 2:

The subject will proceed to the home-monitoring study. Aim of the extended study is to assess sensitivity of seizure detection of sqEEG in comparison to subject's diary in the daily environment, and the tolerability and safety of sqEEG in a period of at least 3 months.

Study protocol of the extended part:

* The subject will be discharged at home after EMU admission with the device and all the necessary information on how to handle it.
* Data on usage times for each participant will be derived from the time stamps and duration of the recorded EEGs as saved by the ELD.
* Adjustment of the anti-seizure medicines will be allowed whenever the clinical conditions will require it. Any changes in the treatment will be noted in the subjects' seizure diary. Data on the use of ASMs will be collected at every study visit.
* Adverse Device Effects (ADEs) will be defined as any unintended or unfavorable response to the system during the study period possibly related to the use of the device or related procedures. ADEs will be classified according to severity based on their impact on daily life as the following: mild (does not interfere with everyday activities), moderate (interferes with some everyday activities), and severe (prevents some everyday activities) (Weisdorf et al., 2019). Serious ADEs will be defined as ADEs requiring hospitalization, leading to death (or would have done so in the absence of treatment) or lasting disability. These definitions will follow the guidance provided in ISO 14155:2011 Clinical investigation of medical devices for human subjects - Good clinical practice.
* Participants will be requested to document all events that they believed to be seizures in a seizure diary. Collection of the time and date will be integrated with the registration of each event. In the paper form, participants have to note time and date by themselves. Participants will be instructed also to provide a seizure description as detailed as possible by using a specific form. Family members or caregivers will be allowed to fill out the seizure description forms. Upon collection, the participants will have the opportunity to comment on the entries to the seizure diary and the seizure descriptions.
* Based on all the information available, self-reported events will be classified following two steps: (1) classification of each event as epileptic or non-epileptic; (2) evaluation of each epileptic seizure and adding a further semiology label as "focal aware seizure (FAS)," "focal impaired awareness seizure (FIAS)," or "uncertain." This distinction will be made by an experienced epileptologist.

At every week after discharge, a review by visual inspection of one week EEG data will be performed, and assessment of the reportability of the sqEEG in comparison to subject's diary, tolerability and safety of the device will be evaluated.

Evaluation of the EEG data by the algorithm for automatic seizure detection will be performed blinded from the results of the visual analysis. In addition, an evaluation of the potential individual clinical impact of the data obtained will be performed.

Visual review of the EEG: a neurophysiology technician trained in reading the sqEEG data will review the raw data from EpiSight (the software for the visualization of sqEEG data, who is part of the device) to identify seizure events blinded from the subject's seizure diary. The detected events will be validated by a supervision of an expert clinical neurophysiologist.

Assessment of tolerability and safety: eventual complaints about tolerability will be collected from the subject and the diary. Side-effects, reported by the subject and in the diary will be analyzed as classified as described above.

Evaluation of the algorithm for automatic seizure detection (ASD): the sqEEG data will be analyzed by the ASD algorithm; the results of the ASD algorithm will be reviewed by investigators blinded from the results of the visual analysis.

Assessment of potential clinical impact: the results of the 3-6 months sqEEG monitoring will be evaluated in terms of their possible impact on patient's management by evaluating its usefulness:

* to evaluate the actual seizure frequency with the ongoing treatment at the time of implantation and compare it with the seizure frequency reported in the diary;
* to prompt of adjustments of the medical treatment and evaluate their effects (the time "before treatment changes" and the time "after treatment changes" should possibly be of comparable length);
* to identify and define patterns of seizure occurrence (circadian occurrence, clustering of seizures) that can be communicated to the subject to eventually counsel him/her on how to behave in the more vulnerable situations;
* in assessing whether support measures (for instance, nocturnal supervision, specialized personnel, safer accommodations) are advised (for example, in cases of seizure frequency being higher than expected in subjects living alone).
* other factors not considered, but suggested by subject or PI to provide a clinical impact.

After 12 weeks of home sqEEG monitoring, subjects will terminate the clinical study and the subscalp electrode is removed. A further follow-up visit will be planned per clinical practice in the months after study termination.

If the doctor and patient judge the device useful an extension study period of other 12 weeks is allowed (to reach 24 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Age > 12 years old, with or without intellectual disabilities;
* Diagnosis of drug resistant seizures, DEE or rare epilepsies ;
* One or more seizure types as established by previous epilepsy history thus allowing to define seizure type and scalp topography of the ictal discharge;
* Availability for the duration of the study (3 months);

Exclusion Criteria:

* Subjects with psychiatric disorders including schizophrenia, bipolar affective disorder, emotionally unstable personality disorder, schizoaffective disorder;
* Subject has skeletal deformities or damage at the proposed implantation site to an extent that impedes correct electrode placement;
* Subject has an infection at implant site;
* Subjects at high risk of surgical complications, such as active systemic infection and hemorrhagic disease;
* Subject has or is exposed to a medical device that delivers electrical energy into the area around the implant (cochlear implant(s));
* Subject has a profession or hobby that includes activity imposing an unacceptable risk for trauma to the device or implant site, e.g. martial arts or boxing;
* Subject has a contraindication to the use of local anesthetic drugs used during implantation- and removal of the device;
* Subject is unable or does not have the necessary assistance to properly operate the device system.
* Pregnancy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the reportability | 12-24 weeks from device activation
  The results (i.e., number of seizures, date and time) will be matched with the subject's seizure diary to look for concordance.

SECONDARY OUTCOMES:
Assessment of Device-Related Adverse Events: | 12-24 weeks from device activation
  Will be collected from the subject during the study visits and by means of a specific form. The presence of the following side-effects will be checked: formation of haematoma or seroma near the implant site; temporary pain, headache, infection and discomfort; skin ischemia potentially inducing necrosis at the implant site due to pressure and compromised local circulation; Infection, swelling, soreness, irritation or itching of the skin at the implant site; occasional headache or pain during long-term use of the device.
Evaluation of the algorithm for automatic seizure detection (ASD) | 12-24 weeks from device activation
  The sqEEG data will be analyzed by the ASD algorithm; the results of the ASD algorithm will be reviewed by investigators blinded from the results of the visual analysis.
Assessment of potential clinical impact | 12 to 24 weeks from device activation
  The results of the 3-month sqEEG monitoring will be evaluated in terms of their possible impact on patient's clinical management

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Meletti, MD, PhD, Principal Investigator — Azienda Ospedaliero Universitaria di Modena - Ospedale Civile di Baggiovara - S.S.D. Neurofisiologia
Locations (4):
- Italy (4):
  - Ospedale pediatrico Bambino Gesù, Roma, Italy
  - Azienda Sanitaria Universitaria Giuliano Isontina, Trieste, Italy
  - S.S.D. Neurofisiologia Clinica - AOU di Modena, Modena, Taly
  - Azienda Ospedaliero Universitaria Federico II - Napoli, Napoli, Taly

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weisdorf S, Gangstad SW, Duun-Henriksen J, Mosholt KSS, Kjaer TW. High similarity between EEG from subcutaneous and proximate scalp electrodes in patients with temporal lobe epilepsy. J Neurophysiol. 2018 Sep 1;120(3):1451-1460. doi: 10.1152/jn.00320.2018. Epub 2018 Jul 11. PMID 29995605
- [Background] Viana PF, Remvig LS, Duun-Henriksen J, Glasstetter M, Dumpelmann M, Nurse ES, Martins IP, Schulze-Bonhage A, Freestone DR, Brinkmann BH, Kjaer TW, Richardson MP. Signal quality and power spectrum analysis of remote ultra long-term subcutaneous EEG. Epilepsia. 2021 Aug;62(8):1820-1828. doi: 10.1111/epi.16969. Epub 2021 Jul 12. PMID 34250608
- [Background] Viana PF, Duun-Henriksen J, Glassteter M, Dumpelmann M, Nurse ES, Martins IP, Dumanis SB, Schulze-Bonhage A, Freestone DR, Brinkmann BH, Richardson MP. 230 days of ultra long-term subcutaneous EEG: seizure cycle analysis and comparison to patient diary. Ann Clin Transl Neurol. 2021 Jan;8(1):288-293. doi: 10.1002/acn3.51261. Epub 2020 Dec 4. PMID 33275838
- [Background] Trivisano M, Specchio N. What are the epileptic encephalopathies? Curr Opin Neurol. 2020 Apr;33(2):179-184. doi: 10.1097/WCO.0000000000000793. PMID 32049741
- [Background] Specchio N, Wirrell EC, Scheffer IE, Nabbout R, Riney K, Samia P, Guerreiro M, Gwer S, Zuberi SM, Wilmshurst JM, Yozawitz E, Pressler R, Hirsch E, Wiebe S, Cross HJ, Perucca E, Moshe SL, Tinuper P, Auvin S. International League Against Epilepsy classification and definition of epilepsy syndromes with onset in childhood: Position paper by the ILAE Task Force on Nosology and Definitions. Epilepsia. 2022 Jun;63(6):1398-1442. doi: 10.1111/epi.17241. Epub 2022 May 3. PMID 35503717
- [Background] Remvig LS, Duun-Henriksen J, Furbass F, Hartmann M, Viana PF, Kappel Overby AM, Weisdorf S, Richardson MP, Beniczky S, Kjaer TW. Detecting temporal lobe seizures in ultra long-term subcutaneous EEG using algorithm-based data reduction. Clin Neurophysiol. 2022 Oct;142:86-93. doi: 10.1016/j.clinph.2022.07.504. Epub 2022 Aug 8. PMID 35987094
- [Background] Pathmanathan J, Kjaer TW, Cole AJ, Delanty N, Surges R, Duun-Henriksen J. Expert Perspective: Who May Benefit Most From the New Ultra Long-Term Subcutaneous EEG Monitoring? Front Neurol. 2022 Jan 20;12:817733. doi: 10.3389/fneur.2021.817733. eCollection 2021. PMID 35126304
- [Background] Kjaer TW, Remvig LS, Helge AW, Duun-Henriksen J. The Individual Ictal Fingerprint: Combining Movement Measures With Ultra Long-Term Subcutaneous EEG in People With Epilepsy. Front Neurol. 2021 Dec 23;12:718329. doi: 10.3389/fneur.2021.718329. eCollection 2021. PMID 35002910
- [Background] Muller AR, Brands MMMG, van de Ven PM, Roes KCB, Cornel MC, van Karnebeek CDM, Wijburg FA, Daams JG, Boot E, van Eeghen AM. Systematic Review of N-of-1 Studies in Rare Genetic Neurodevelopmental Disorders: The Power of 1. Neurology. 2021 Mar 16;96(11):529-540. doi: 10.1212/WNL.0000000000011597. Epub 2021 Jan 27. PMID 33504638
- [Background] Elger CE, Hoppe C. Diagnostic challenges in epilepsy: seizure under-reporting and seizure detection. Lancet Neurol. 2018 Mar;17(3):279-288. doi: 10.1016/S1474-4422(18)30038-3. PMID 29452687
- [Background] Cook MJ, O'Brien TJ, Berkovic SF, Murphy M, Morokoff A, Fabinyi G, D'Souza W, Yerra R, Archer J, Litewka L, Hosking S, Lightfoot P, Ruedebusch V, Sheffield WD, Snyder D, Leyde K, Himes D. Prediction of seizure likelihood with a long-term, implanted seizure advisory system in patients with drug-resistant epilepsy: a first-in-man study. Lancet Neurol. 2013 Jun;12(6):563-71. doi: 10.1016/S1474-4422(13)70075-9. Epub 2013 May 2. PMID 23642342
- [Background] Blachut B, Hoppe C, Surges R, Elger C, Helmstaedter C. Subjective seizure counts by epilepsy clinical drug trial participants are not reliable. Epilepsy Behav. 2017 Feb;67:122-127. doi: 10.1016/j.yebeh.2016.10.036. Epub 2017 Jan 28. PMID 28139449
- [Background] Blachut B, Hoppe C, Surges R, Stahl J, Elger CE, Helmstaedter C. Counting seizures: The primary outcome measure in epileptology from the patients' perspective. Seizure. 2015 Jul;29:97-103. doi: 10.1016/j.seizure.2015.03.004. Epub 2015 Apr 13. PMID 26076850